CLINICAL TRIAL: NCT05010902
Title: Pregnancy Cohort in Multiple Sclerosis (MS)
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Nadja Siebert, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: PreCoMS
Record Dates: First submitted 2021-07-21; First posted 2021-08-18 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis (MS); Clinically Isolated Syndrome (CIS)
Keywords: Pregnancy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis: Patients with clinically isolated syndrome, relapsing-remitting or progressive multiple sclerosis

SUMMARY:
Multiple sclerosis (MS) is a common inflammatory demyelinating disorder of the central nervous system frequently affecting females in their reproductive phase of life. In this prospective observational study, we obtain data on the outcome of pregnancies in MS patients and the influence of pregnancy on clinical, laboratory and MRI parameters in MS.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* signed informed consent
* diagnosis of multiple sclerosis or clinically isolated syndrome

Exclusion Criteria:

* clinically relevant comorbidities
* contraindications for MRI, e.g. pacemaker, metal implants, allergy against gadolinium
* alcohol or drug abuse

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruted at neurological outpatient clinics and neurological clinics of the Charité and neurologists' medical practices.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time until relapse | 12 months after delivery compared to baseline
  Time (in days) until relapse during the observation period

SECONDARY OUTCOMES:
Number of T2 lesions | 12 months after delivery compared to baseline
  Number of T2 lesions in spinal and cerebral magnetic resonance imaging
Number of gadolinium enhancing lesions | 12 months after delivery compared to baseline
  Number of gadolinium enhancing lesions in spinal and cerebral magnetic resonance imaging
Volume of T2 lesions | 12 months after delivery compared to baseline
  Volume of T2 lesions in spinal and cerebral magnetic resonance imaging
Volume of gadolinium enhancing lesions | 12 months after delivery compared to baseline
  Volume of gadolinium enhancing lesions in spinal and cerebral magnetic resonance imaging
Change in immune cell phenotypes | 12 months after delivery compared to baseline
  Change in immune cell phenotypes of peripheral blood mononuclear cells (PBMC)
Galectin-1 | 12 months after delivery compared to baseline
  Change in serum galectin-1 concentration measured by ELISA
Galectin-3 | 12 months after delivery compared to baseline
  Change in serum galectin-3 concentration measured by ELISA
Galectin-9 | 12 months after delivery compared to baseline
  Change in serum galectin-9 concentration measured by ELISA
Neurofilament (NfL) | 12 months after delivery compared to baseline
  Change in neurofilament serum concentration by using Simoa NfL assay
Pro-inflammatory interleukin-17 | 12 months after delivery compared to baseline
  Change in interleukin-17 serum concentration assessed by ELISA
Anti-inflammatory interleukin-10 | 12 months after delivery compared to baseline
  Change in anti-inflammatory interleukin-10 serum concentration assessed by ELISA
Autoantibody profiling | 12 months after delivery compared to baseline
  Identification and quantification of autoantibodies by using protein microarray and ELISA
Fecal microbiome composition | 12 months after delivery compared to baseline
  Composition of fecal microbiome measured by 16S Sequencing
Thickness of the retinal nerve fibre layer | 12 months after delivery (compared to baseline)
  Thickness of the retinal nerve fibre layer by Optical Coherence Tomography (OCT)
Total macular volume (TMV) | 12 months after delivery compared to baseline
  Total macular volume by Optical Coherence Tomography (OCT)
Mini-International Neuropsychiatric Interview (M.I.N.I.) German Version 5.0.0 Module A-C | 12 months after delivery compared to baseline
  Structured diagnostic interview to assess depression, dysthymia and suicidality
Montgomery-Asberg Depression Rating Scale (MADRS) | 12 months after delivery compared to baseline
  Rating of ten depression related symptoms on a scale from 0 to 6 (higher numbers indicate more severe symptoms)
Beck Depression Inventory (BDI-II) | 12 months after delivery compared to baseline
  Rating of 21 depression related symptoms on a scale from 0 to 3 (higher numbers indicate more severe symptoms)
Edinburgh Postpartum Depression Scale (EPDS) | 12 months after delivery compared to baseline
  Self-report survey containing 10 items, each item is rated 0-3 (higher scores indicate a higher probability of postpartum depression)
Modified Fatigue Inventory Scale (MFIS) | 12 months after delivery compared to baseline
  Self-report survey containing 21 items, each item is rated 0-4 (higher scores indicate a greater impact of fatigue on a person's activities)
Fatigue Severity Scale (FSS) | 12 months after delivery compared to baseline
  A self-report survey consisting of 11 items, each item ranges from 1 to 7 (higher scores indicate higher levels of fatigue)
Visual Fatigue Analogue Scale (VFAS) | 12 months after delivery compared to baseline
  A self-administered, single scale indication measuring visual fatigue, ranging from 0 to 100 (higher scores indicate worse fatigue)
Short-Form Health Survey (SF-36) | 12 months after delivery compared to baseline
  A self-report survey measuring health in eight dimensions (higher scores indicate less disability)

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Siebert, MD, Principal Investigator — Experimental & Clinical Research Unit, Charité Universitätsmedizin Berlin
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal